CLINICAL TRIAL: NCT05532839
Title: Effects of Self-paced High-intensity Interval Training and Moderate Intensity Continuous Training on the Physical Performance and Psychophysiological Responses in Recreationally Active Young Adults
Brief Title: Self-paced High-intensity Interval Training and Moderate Intensity Continuous Training in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0415
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Psychophysiologic Reaction
Keywords: High intensity interval training; Moderate intensity continuous training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): High-intensity interval training is a training that cycles between high bursts of activity and predetermined times of less intensive exercise or rest period.
  Interventions: Other: High intensity interval training
- Moderate intensity continuous interval training (Experimental): Moderate-intensity continuous training consists of periods followed by 50 minutes of exercise - bicycling, running, jogging, marching, paddling, etc. - at a recorded frequency of 70-75 percent maximal heart rate.
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: High intensity interval training — The therapy lasted 6 weeks, and HIIT comprised of two 12-24 × 30 second high-intensity runs separated by thirty seconds of relaxation.
  Arms: High intensity interval training
Other: Moderate intensity continuous training — The MICT ran continuously for 24-48 minutes. From the day of the six weeks intervention strategies, the mentioned assays were conducted: Yo-Yo Intermittent Recovery Test level 1, repeated sprint ability , sprint test, alter of way test which is t drill, and physical activity enjoyment scale and shuttle run. Through these trainings, individuals in both groups must follow the old their balanced meal.
  Arms: Moderate intensity continuous interval training

SUMMARY:
Study will be randomized clinical trial. Data will be collected from non probability convenient sampling technique. Total 26 participants from Pakistan Sports Board will be selected and randomly allocated in two different groups i.e. Group A and Group B. Group A will be given high intensity interval training and Group B will be on moderate intensity continuous training. Statistical package for the social sciences will be used to analyze the results by using parametric test after confirming normality of data.

DETAILED DESCRIPTION:
Recreational activities are those in which you genuinely engage with others to have fun and relax in your leisure time. This includes activities that require physical activity as well as connections and play with others. They are not activities that you can finish totally on your alone; while you can try to do some with your own, you will miss out on the enjoyment of doing that with others

High-intensity interval training is a training that cycles between high bursts of activity and predetermined times of less intensive exercise or rest period. The therapy lasted 6 weeks, and HIIT comprised of two 12-24 × 30 second high-intensity runs separated by thirty seconds of relaxation.

Moderate-intensity continuous training consists of periods followed by 50 minutes of exercise- bicycling, running, jogging, marching, paddling, etc. - at a recorded frequency of 70-75 percent maximal heart rate. The MICT ran continuously for 24-48 minutes. From the day of the six weeks intervention strategies, the mentioned assays were conducted: Yo-Yo Intermittent Recovery Test level 1, repeated sprint ability , sprint test, alter of way test which is t drill, and physical activity enjoyment scale and shuttle run. Through these trainings, individuals in both groups must follow the old their balanced meal.

ELIGIBILITY:
Inclusion Criteria:

* Both genders was included in our study.
* Participants of age of 16 to 35 years were included.
* Included those participants who were playing sports such as cricket, football, basketball and tennis and their training workload of less than three training units per week and less than one eight minutes, also doing core strength training, also doing cardio trainings and group exercise, from the last two years.

Exclusion Criteria:

* Adults who were having history of any trauma from last 6 month were excluded.
* SOB or any other cardiopulmonary disease.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Yo-Yo Intermittent Recovery Test level 1 (YYIRTL-1) | 3 months
  To assess an athlete's capacity to undertake high-intensity aerobic activities continuously
Repeated sprint ability (RSA) | 3 months
  Sprint test of 10-30 meters to improve and uphold maximal exertion through consecutive sprints
Change of direction test (T-drill) | 3 months
  It includes forward, sideways, and revers movements
Training rating of perceived exertion (RPE) | 3 months
  It is based on the physical experiences a human has during physical exercise, such as elevated heart rate, increase breathing or respiratory rate, increased perspiration, and muscular tiredness.
Physical activity enjoyment scale (PACES) | 3 months
  It is an 18-item scale that examines physical activity pleasure by simply asking to score "how you feel right here about the physical activity you've been performing
Shuttle run test (PACER) | 3 months
  The thirty feet agility Shuttle Run is indeed an agility assessment wherein the opponent sprints switch between different line segments as rapidly as feasible, trying to pick up wooden blocks for a distance travelled of 8 m. main goal: this is a way of measuring of power and speed

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Sadia Afzaal Sukhera, Lahore, Lahore, Punjab, Pakistan, Pakistan